CLINICAL TRIAL: NCT00373620
Title: A Phase II Trial of Radiation Therapy With Concurrent Paclitaxel Chemotherapy in High-Risk Endometrial Cancer Patients After Operation.
Brief Title: A Safety and Efficacy of CCRT With Paclitaxel as Adjuvant Therapy to Post-Operative Advanced Endometrial Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korean Gynecologic Oncology Group (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KGOG2001
Record Dates: First submitted 2006-09-06; First posted 2006-09-08 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2005-12

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; high risk; weekly paclitaxel; Cuncurrent chemoradiation
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Paclitaxel

INTERVENTIONS:
Drug: paclitaxel

SUMMARY:
The purpose of this study is to determine whether post-operative concurrent chemoradiation with paclitaxel is effective and safe in the treatment of high risk postoperative endometrial cancer patients.

DETAILED DESCRIPTION:
Postoperative radiotherapy (RT) is the most used adjuvant treatment in high risk endometrial cancer (HREC), and it appears to reduce the incidence of pelvic relapses but doesn't seem to improve survival. Paclitaxel (P) has shown in vitro and clinical activity against endometrial cancer, and it is also a potent radiosensitizer by blocking dividing cells in G2/M phase. This study is to evaluate the efficacy and safety of a treatment with concomitant weekly chemotherapy with paclitaxel and RT in high risk advanced endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients undertaken total hysterectomy, bilateral salpingoophorectomy, washing cytology, pelvic and paraaortic lymph node dissection
* Patients must have the diagnosis of endometrioid type adenocarcinoma with stage III, IV.
* Patients must have a GOG performance of 0, 1, or 2.
* Patients must have expected life span over 6 months.

Exclusion Criteria:

* Patients with peripheral neurotoxicity over grade 2 in CTC criteria.
* Patients with history of chemotherapy or radiation treatment.
* patients with history of arrhythmia,congestive heart failure.
* Patients with intractable infection.

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-01

PRIMARY OUTCOMES:
Two year progression free survival

SECONDARY OUTCOMES:
toxicity profile

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Hoon Kim, Professor, Study Chair — Yong-Dong Severance Hospital
Locations (1):
- Young-Dong Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Cho H, Nam BH, Kim SM, Cho CH, Kim BG, Ryu HS, Kang SB, Kim JH. A phase 2 trial of radiation therapy with concurrent paclitaxel chemotherapy after surgery in patients with high-risk endometrial cancer: a Korean Gynecologic Oncologic Group study. Int J Radiat Oncol Biol Phys. 2014 Sep 1;90(1):140-6. doi: 10.1016/j.ijrobp.2014.05.024. Epub 2014 Jul 8. PMID 25015202